CLINICAL TRIAL: NCT06300723
Title: Clinical Study to Evaluate the Safety and Efficacy of Single Dose Intravenous Infusion of CRISPR/Cas9-edited Autologous CD34 + Hematopoietic Stem/Progenitor Cells (BRL-101) in the Treatment of Severe Sickle Cell Disease
Brief Title: Clinical Study of BRL-101 in Severe SCD
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: Bioray Laboratories (Industry)
Collaborators: First Affiliated Hospital of Guangxi Medical University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2024-BRL-101-SCD-01
Record Dates: First submitted 2024-03-03; First posted 2024-03-08 (Actual); Last update posted 2024-07-31 (Actual); Status verified 2024-05

CONDITIONS: Sickle Cell Disease
MeSH Terms: conditions — Anemia, Sickle Cell

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- BRL-101 (Experimental): Autologous CD34+ hHSPCs modified with CRISPR-Cas9 at the BCL11A gene. Subjects will receive a single infusion of BRL-101.
  Interventions: Drug: BRL-101

INTERVENTIONS:
Drug: BRL-101 — CD34 + autologous hematopoietic stem and progenitor cells edited at the BCL11A gene.
  Other Names: Autologous hematopoietic stem and progenitor cells injection

SUMMARY:
This is a single center, non-randomized, open label, single-dose study in subjects with Sickle Cell Disease (SCD). The study will evaluate the safety and efficacy of autologous CRISPR-Cas9 modified CD34+ human hematopoietic stem and progenitor cells (hHSPCs) (BRL-101).

DETAILED DESCRIPTION:
This clinical trial is a single-arm, single-dose, single center, open-label study without dose escalation. The primary objective is to explore the safety of the study drug in SCD. Myeloablative conditioning and administration for the remaining subjects can only be started after the first subject completes dosing and safety observation and assessment.

ELIGIBILITY:
Inclusion Criteria:

-

Subjects must meet all the following inclusion criteria to be eligible for enrolment into the study:

1. Subject (or their legally authorized representative or guardian) will sign and date an informed consent form (ICF) and, where applicable, an assent form.
2. Subjects 3 to 35 years of age, inclusive, on the date of informed consent.
3. Clinically confirmed severe SCD, genotypes include: βS/βS, βS/β + or βS/β0. Severe SCD is defined as having at least 2 VOC events per year during the 2 years prior to screening and requiring appropriate supportive care, including a pain management program, HU therapy (if indicated).
4. Karnofsky performance status of ≥80% for subjects ≥16 years of age. Lansky performance status of ≥80% for subjects <16 years of age (see Appendix 1 and 2).
5. Eligible for autologous stem cell transplant as per investigator's judgment.
6. Willing and able to comply with scheduled visits, treatment plan, laboratory tests, contraceptive guidelines, and other study procedures.
7. Willing to participate in an additional long-term follow-up study after completion of this study .
8. Subjects of childbearing potential must use effective contraception for at least 6 months after BRL-101 infusion during the study.

Exclusion Criteria:

-

Subjects meeting any of the following criteria are not eligible for enrolment in the study:

1. Known contraindications, intolerance, or hypersensitivity to hematopoietic stem cell mobilizers, busulfan injection, or dimethyl sulfoxide (DMSO) or study drug-related components.
2. Eligible for allogeneic hematopoietic stem cell transplantation and have found HLA-identical donors.
3. Prior allo-HSCT, gene therapy or gene editing therapy.
4. Clinically significant and active bacterial, viral, fungal, or parasitic infection as determined by the investigator.
5. HbF level >15.0%, irrespective of concomitant treatment with HbF inducing treatments such as HU.
6. Treatment with regular RBC transfusions that, in the opinion of the investigator, cannot be interrupted after engraftment.
7. More than 10 unplanned hospitalizations or emergency department visits related to SCD in the 1 year before screening and the investigator considered this to be a significant chronic pain rather than an acute pain crisis.
8. A history of clinically significant transcranial Doppler (TCD) test abnormalities or test abnormalities in the opinion of the investigator.
9. History of untreated Moyamoya disease or presence of Moyamoya disease at Screening that in the opinion of the investigator puts the subjects at the risk of bleeding.
10. the subject has participated in other clinical studies and used drugs within 3 months before screening.
11. White blood cell count < 3 × 109/L and/or platelet count < 100 × 109/L not due to hypersplenism as judged by the investigator.
12. INR > 1.5×ULN, APTT > 1.5×ULN.
13. Creatinine > 1.5 × ULN or endogenous creatinine clearance < 60 ml/min (calculated according to the Cockcroft-Gault formula, see Appendix 3).
14. ALT or AST> 3×ULN, or direct bilirubin value > 2.5×ULN.
15. Severe iron overload with serum ferritin ≥ 5000 ng/ml, liver iron > 15 mg Fe/g dry weight (or liver MRIT2* < 1.4 ms or > 588 Hz), or heart MRI-T2* < 10 ms.
16. LVEF < 50%.
17. DLco < 50% predicted (corrected haemoglobin or/and alveolar volume) or forced vital capacity (FVC) (measured/predicted) < 60% (For children for whom DLco could not be determined), or abnormal blood gas analysis (for younger children with undetectable ventilatory function only).
18. Hepatitis B virus surface antigen (HBsAg) positive or HBV-DNA positive; hepatitis C virus (HCV) antibody positive; human immunodeficiency virus (HIV) antibody positive; syphilis (TP) -specific antibody positive; Epstein-Barr virus EBV-DNA positive; cytomegalovirus CMV-DNA positive.
19. History of a significant bleeding disorder.
20. History or family history of malignancy or myeloproliferative disorder.
21. Any prior or current cardiovascular system diseases, such as congestive heart failure, arrhythmia, myocardial disease, valvular heart disease or pulmonary hypertension; cirrhosis, liver fibrosis or active hepatitis; central nervous system diseases or mental illness.
22. Presence of immune dysfunction or endocrine disorders, such as insulin-dependent diabetes mellitus, hyperthyroidism, or insufficiency.
23. Pregnant or breastfeeding females.
24. Any condition that, in the opinion of the investigator, would make participation in this clinical study inappropriate.

Ages: 3 Years to 35 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 3 (Estimated)
Dates: Start 2024-07-29 (Actual); Primary Completion 2026-03-20 (Estimated); Study Completion 2026-06-15 (Estimated)

PRIMARY OUTCOMES:
Proportion of stem cell engrafted subjects | Within 42 Days After BRL-101 Infusion
  Stem cell engraftment was defined as an absolute peripheral blood neutrophil count of ≥ 0.5 × 109/L for 3 consecutive days following BRL-101 intravenous infusion
Time to neutrophil engraftment | Within 42 Days After BRL-101 Infusion
  Defined as Day 1 of absolute peripheral blood neutrophil count ≥ 0.5 × 109/L for 3 consecutive days
Frequency, severity, and relationship to BRL-101 of adverse events over 12 months following BRL-101 infusion | Up to 12 Months After BRL-101 Infusion
  Adverse events assessed according to NCI-CTCAE v5.0 criteria

CONTACTS AND LOCATIONS:
Overall Officials: Yongrong Lai, phD, Study Chair — First Affiliated Hospital of Guangxi Medical University
Locations (1):
- First Affiliated Hospital of Guangxi Medical University, Nanning, Guangxi, China

IPD SHARING:
Plan to Share IPD: No